CLINICAL TRIAL: NCT05624008
Title: Clinical Performance of Bioactive Bioceramic Glass Ionomer Restorations vs Conventional High Viscous Glass Ionomer Restorations in Geriatric Patients With Carious Cervical Lesions: A One Year Randomized Clinical Trial.
Brief Title: Clinical Performance of Bioceramic vs High Viscosity GIC for Cervical Restorations of Geriatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Mohammed Abd Al-Naieem, Master degree candidate, Conservative Dentistry Department, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bioceramic GIC
Record Dates: First submitted 2022-11-05; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Cervical Caries
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioceramic glass ionomer restoration (Experimental): Calcium aluminate modified glass ionomer
  Interventions: Other: Bioceramic glass ionomer restoration
- Resin modified glass ionomer restoration (Active Comparator): type II resin modified glass ionomer cement
  Interventions: Other: Resin modified glass ionomer restoration

INTERVENTIONS:
Other: Bioceramic glass ionomer restoration — bioactive glass ionomer with unique biocompatibility and biological regenerative properties
  Arms: Bioceramic glass ionomer restoration
Other: Resin modified glass ionomer restoration — A hybrid of glass ionomer and composite resin with acid-base and polymerizable components
  Arms: Resin modified glass ionomer restoration

SUMMARY:
The aim of this study is to clinically evaluate the performance of the bioceramic glass ionomer compared to conventional high viscosity glass ionomer for restoration of carious cervical lesions in geriatric patients over 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric patients aged above 55 years
* Patients with untreated carious lesions
* Patients who have at least 20 teeth under occlusion
* Patients with normal occlusion
* Vital teeth with carious cervical lesion with asymptomatic vital pulp.
* Teeth with no or minimum mobility.
* Teeth with normal occlusion.
* Teeth with surrounding healthy gingiva and supporting-structures.

Exclusion Criteria:

* Patients who are unable to return for recall appointments
* Presence of abnormal oral, medical or mental conditions.
* Patients with severe medical diseases.
* Patients with xerostomia
* Patients with parafunctional habits.
* Non vital teeth.
* Teeth with signs or symptoms of pulpitis.
* Teeth with non carious lesions.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change in Marginal adaptation score | Baseline, 3 months, 6 months, 12 months
  Modified USPHS criteria with Alpha, Bravo and Charlie scores (Categorical)

SECONDARY OUTCOMES:
Change in Retention score | Baseline, 3 months, 6 months, 12 months
  Modified USPHS criteria with Alpha, Bravo and Charlie scores (Categorical)
Change in Color match score | Baseline, 3 months, 6 months, 12 months
  Modified USPHS criteria with Alpha, Bravo and Charlie scores (Categorical)
Change in Marginal discoloration score | Baseline, 3 months, 6 months, 12 months
  Modified USPHS criteria with Alpha, Bravo and Charlie scores (Categorical)
Change in Secondary caries score | Baseline, 3 months, 6 months, 12 months
  Modified USPHS criteria with Alpha, Bravo and Charlie scores (Categorical)
Change in Wear score | Baseline, 3 months, 6 months, 12 months
  Modified USPHS criteria with Alpha, Bravo and Charlie scores (Categorical)
Change in Postoperative hypersensitivity score | Baseline, 3 months, 6 months, 12 months
  Modified USPHS criteria with Alpha, Bravo and Charlie scores (Categorical)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, ElManial, Egypt

IPD SHARING:
Plan to Share IPD: No